CLINICAL TRIAL: NCT02833649
Title: Comparative Analysis of the Visual Performance in Patients With Stable Keratoconus After Implantation of the Toric Implantable Collamer Lens (TICL).
Brief Title: Comparative Analysis of the Visual Performance After TICL Implantation in Patients With Stable Keratoconus
Acronym: TICL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Farideh Doroodgar, Clinical Professor, Shahid Beheshti University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShaheedBU
Record Dates: First submitted 2016-07-04; First posted 2016-07-14 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Keratoconus
Keywords: Keratoconus; Crosslinking; Toric ICL
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Toric Implantable contact Lens (Experimental): The Visian implantable collamer lens (Staar Surgical AG, Nidau, Switzerland), is a monoblock single-piece plate haptic lens made of collamer (an extremely hydrophilic and highly biocompatible flexible collagen copolymer with a refractive index of 1.452 that is permeable to oxygen and nutrients
  Interventions: Device: Toric Implantable collamer Lens

INTERVENTIONS:
Device: Toric Implantable collamer Lens — The toric implantable collamer lens (TICL) is conventionally indicated for the Correcting the refractive error in keratoconus using the TICL is an off label use of the lens.
  Other Names: TICL

SUMMARY:
To report on 4-year postoperative safety, efficacy, stability and predictability outcomes(to evaluate the visual, refractive, contrast sensitivity, defocus curve and aberrometric data preoperation, and compare with a similar postoperative outcomes) with the Toric Implantable Contact Lens (TICL) for Stable keratoconus. Investigators will study the four-year follow-up from this standardized, multi-center clinical investigation, support from clinical and optical viewpoints TICL implantation, in stable keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* age (25-38).
* Stable refraction was distinctive by 6 subjective refractions within ± 0.50 diopters(D) of spherical equivalent during 6 months after CXL.
* best spectacle-corrected visual acuity (BCVA) of +0.4 LogMAR (20/40) or better, -clear central cornea.
* normal anterior chamber depth at least 3 mm to endothelium .
* intraocular pressure (IOP)<20 mm Hg and preoperative endothelial cell count related to age and the anterior chamber depth with regard to Food and Drug Administration recommendations.
* Width of Angle greater than 30°, a pupil diameter of less than 6.25 mm.

Exclusion Criteria:

* Patients with central corneal thickness of less than 450 μm.
* endothelial cell count of less than 2,000 cells/mm2 .
* anterior chamber depth of <3 mm from endothelium to anterior capsule .
* Corneal opacification or scars, cataract, retinal detachment, glaucoma, retinopathy, macular degeneration, neuro ophthalmic diseases or ocular inflammation, history of keratitis (any form), peripheral marginal degeneration, previous corneal and/or intraocular surgeries, and autoimmune and/or connective tissue disease. The central corneal thickness limit of 450 μm would account for around 400 μm of remaining stromal thickness after removal of the epithelium, which is considered as the safety thickness for the residual stroma to avoid endothelial cell damage during the CXL procedure.

Ages: 25 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity (UCVA,BCVA) by Snellen chart | Up to 4 years after surgery

SECONDARY OUTCOMES:
Refractive error by Auto Kerato-Refractometer | Until 4 years after surgery
Defocus curve by Phoropter | Up to 4 years after surgery
Patient satisfaction to measure the patients' subjective assessment of visual improvement by a validated questionnaire | up to 4 years after surgery
Contrast sensitivity by MediWorks C901 Acuity Chart (Shanghai MediWorks Precision Instruments Co, Ltd, Shanghai, China. | up to 4 years after surgery
Aberrometry by Ray Tracing | Up to 4 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Farideh Doroodgar, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doroodgar F, Niazi F, Sanginabadi A, Niazi S, Baradaran-Rafii A, Alinia C, Azargashb E, Ghoreishi M. Comparative analysis of the visual performance after implantation of the toric implantable collamer lens in stable keratoconus: a 4-year follow-up after sequential procedure (CXL+TICL implantation). BMJ Open Ophthalmol. 2017 Sep 28;2(1):e000090. doi: 10.1136/bmjophth-2017-000090. eCollection 2017. PMID 29354720